CLINICAL TRIAL: NCT05548647
Title: Short- and Long-term Effects of Once Weekly Semaglutide 2.4 mg on Appetite, Eating Behavior, and Psychosocial Status
Brief Title: Semaglutide Treatment, Appetite, and Eating Behavior: Long-term Effects
Acronym: STABLE Wt Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 850370
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Semaglutide; Body weight; Obesity; weight loss; medication; overweight; lifestyle modification; diet; exercise; Body Weight Changes; Appetitive Behavior
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss; Overweight; Motor Activity; Body Weight Changes; Appetitive Behavior | interventions — Behavior Therapy; Dosage Forms; semaglutide

STUDY DESIGN:
Intervention Model Description: Study 1 is a double-blind, placebo-controlled, randomized controlled, long-term treatment trial. Study 2 is a double-blind, medication withdrawal trial, re-randomized treatment trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Treatment + Placebo (Active Comparator): Behavioral treatment (lifestyle modification counseling for weight loss) plus placebo
  Interventions: Behavioral: Behavioral Treatment; Drug: Placebo
- Behavioral Treatment + Medication (Active Comparator): Behavioral treatment (lifestyle modification counseling for weight loss) plus semaglutide
  Interventions: Behavioral: Behavioral Treatment; Drug: Semaglutide 2.4 MG/0.75 ML Subcutaneous Solution [WEGOVY]

INTERVENTIONS:
Behavioral: Behavioral Treatment — All participants, regardless of medication assignment, will receive the same 60-week behavioral weight loss program. Brief (15-minute), individual lifestyle counseling sessions will be delivered by a psychologist, behavioral health counselor, or registered dietitian (or other trained health care provider) at weeks 0 (i.e., baseline/randomization), 2, 4 and every fourth week from week 4 to week 60 (17 sessions) of Study 1. Subjects will be instructed to consume a self-selected diet of 1200-1500 kcal/day (for those who weigh < 250 lb) or 1500-1800 kcal/day (for those who weigh ≥250 lb). They will be instructed to engage in low-to-moderate intensity physical activity (e.g., walking), gradually building to a goal of ≥150 minutes per week (spread across 5 days) by week 40. They will be instructed to use calorie counting and self-monitoring to meet their goals.
  Other Names: Lifestyle modification; Behavioral weight loss; Lifestyle intervention
Drug: Placebo — An inactive saline solution administered via subcutaneous injection
  Other Names: Placebo for medication
  Arms: Behavioral Treatment + Placebo
Drug: Semaglutide 2.4 MG/0.75 ML Subcutaneous Solution [WEGOVY] — Semaglutide 2.4 mg is a once weekly subcutaneous glucagon-like peptide-1 (GLP-1) receptor agonist that has been FDA approved for weight loss
  Other Names: Wegovy
  Arms: Behavioral Treatment + Medication

SUMMARY:
This study will evaluate the effect of semaglutide on eating behavior, appetite (hunger/fullness), and food liking in the long-term, as compared to placebo. All participants will receive lifestyle modification (diet and exercise) counseling, and will be prescribed the FDA-approved weight loss medication, semaglutide, or placebo (an inactive saline solution) for 72 weeks.

DETAILED DESCRIPTION:
This trial consists of a single 72-week treatment period during which two studies will be conducted. Study 1 (i.e., long-term treatment trial; weeks 0-60) is a 60-week, single center, double-blinded, randomized controlled, parallel group design trial, and Study 2 (i.e., re-randomized medication withdrawal trial; weeks 60-72) is a separate, 12-week, double-blind, re-randomized medication withdrawal trial.

The long-term treatment trial (Study 1) will randomly assign (in a 3:2 semaglutide:placebo ratio) 120 subjects with a body mass index (BMI) ≥30 kg/m2, or ≥27 kg/m2 with ≥1 obesity-related co-morbidities, to 60 weeks of: 1) placebo with moderate intensity lifestyle intervention (as used in STEP 1); or 2) semaglutide 2.4 mg with the same lifestyle intervention. All subjects will receive 60 weeks of trial product, which will be up-titrated over 16 weeks in those assigned to semaglutide 2.4 mg. They will complete assessments of energy intake, appetite, food reward, mood, symptoms of disordered eating, and anthropomorphic measurements at baseline (week 0) and weeks 20, 40, and 60.

The primary aim in the initial long-term treatment trial will be to compare the long-term effect of semaglutide 2.4 mg vs placebo on ad libitum energy intake during a lunch meal at weeks 20, 40, and 60. Confirmatory secondary aims will test the effect of semaglutide 2.4 mg at weeks 20, 40 and 60 on subjective appetite ratings (both measured during a standardized breakfast in the lab and as experienced more globally over the past week), explicit food reward, as measured with the Power of Food Scale (24), and implicit food reward, as measured with the Leeds Food Preference Task (25, 26). Measures of food cravings, mood, eating disorder symptoms, and self-report measures of eating behavior will be considered supportive secondary endpoints and will provide additional evidence of the medication's safety and efficacy.

Following the completion of Study 1 at week 60, all subjects who complete a week 60 assessment and remain on drug will be enrolled in Study 2. Semaglutide-treated subjects will be re-randomized (in a 1:4 semaglutide:placebo ratio) to receive semaglutide 2.4 mg or placebo for 12 weeks. All subjects originally assigned to placebo will continue with that medication for an additional 12 weeks. Both researchers and subjects will remain blinded to subjects' original and re-randomized (or continued) treatment assignments. The goal of this re-randomized medication withdrawal period will be to compare the 80% of subjects originally assigned to semaglutide 2.4 mg who receive placebo at week 60 (semaglutide-to-placebo group) to the subjects originally randomized to placebo (continuous-placebo group) on all primary and secondary outcome measures at week 72 (after controlling for Study 1 baseline/week 0 values). All subjects will terminate trial product at cumulative week 72 and will return to clinic for a final safety visit at week 76.

Outcome assessments including ad libitum energy intake, subjective measures of appetite, food reward, eating behavior, mood, and eating disorder symptoms will occur at weeks 0, 20, 40, and 60 of Study 1 and at week 12 (72 weeks from original randomization) of the re-randomized treatment period. Measurements of body weight, waist circumference, blood pressure, pulse, and global, past-week appetite and food cravings (COEQ) also will be collected every 4 weeks throughout both treatment studies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who report a desire to lose weight
2. Aged 18-70 years
3. Body mass index [BMI] ≥ 30 kg/m2 or BMI ≥ 27 kg/m2 with an obesity-related comorbidity (e.g., treated or untreated hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease)
4. Eligible female patients will be:

   * non-pregnant, evidenced by a negative urine pregnancy test
   * non-lactating
   * surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study
5. Subjects must

   * Plan to remain in the Philadelphia area for the next 1.5 years.
   * Ability to provide informed consent before any trial-related activities.

Exclusion Criteria:

1. A diagnosis of type I or II diabetes
2. Hemoglobin A1c (HbA1c) > 6.5%
3. Uncontrolled hypertension (blood pressure ≥ 160/100 mm Hg)
4. Clinically significant hepatic (i.e., liver fibrosis, cirrhosis or confirmed NASH) or renal disease
5. Uncontrolled thyroid disease
6. Experienced a cardiovascular event (e.g., stroke, myocardial infarction) in the last 6 months, congestive heart failure, or heart block greater than first degree
7. A history of acute pancreatitis in the last 6 months
8. Any history of chronic pancreatitis
9. A history of malignancy (other than non-melanoma skin cancer) within the last 5 years
10. A personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2
11. A self-reported change in body weight >5kg (11 lbs) within 90 days before screening
12. Used within the last 6 months medications known to produce weight loss/gain (e.g., medications approved for weight loss, oral steroids, antipsychotic medications) or any GLP-1 receptor agonist.
13. Known or suspected allergy or hypersensitivity to trial medication(s), excipients, or related products
14. The receipt of any investigational drug within 6 months prior to this trial
15. Applicants with current severe major depressive disorder (BDI-II score ≥ 29 or Patient Health Questionnaire-9 [PHQ-9] score > 15) or severe anxiety disorder
16. Applicants with current, active suicidal ideation, and/or a suicide attempt within the past year (such individuals will be referred for psychiatric treatment if they have not previously received it).
17. Any severity of psychotic or bipolar disorder
18. Bulimia nervosa diagnosis within the past 5 years
19. Self-reported alcohol or substance abuse within the past 6 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
20. History of (or plans to receive in the next 1.5 years) bariatric surgery or a weight loss device. (However, the following will be allowed: liposuction or abdominoplasty > 1 year before screening, laparoscopic banding if removed > 1 year before screening, intragastric balloon or aspire assist if removed > 1 year before screening.)
21. Inability to walk 5 blocks or more (comfortably) or engage in another form of aerobic activity.
22. Women who are nursing, pregnant, or planning to become pregnant in the next 1.5 years or are not using adequate contraceptive measures
23. Previous participation in this trial (e.g., randomized but failed to participate)
24. Changes to any chronic medication (type or dosage) within the past 3 months.
25. Food allergy or dietary preference that would prevent the individual from consuming the standard breakfast or ad libitum lunch.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake (kcal) during a buffet lunch meal (4 hrs after standardized breakfast) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Primary outcome

SECONDARY OUTCOMES:
Laboratory-based appetite measured as a composite of visual analogue scale ratings (hunger, fullness, satiety, prospective consumption) when fasting and after eating (area under the curve). This is a single outcome calculated by combining the VAS ratings | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Secondary confirmatory outcome
Global subjective appetite (e.g., hunger, fullness, food preoccupation) over the past week measured using the Control of Eating Questionnaire (COEQ) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Secondary confirmatory outcome
Explicit responsiveness to the food environment measured by the summary score of the Power of Food Scale (15-item version) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Secondary confirmatory outcome
Implicit food wanting of high-fat, savory foods measured using the Leeds Food Preference Task | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Secondary confirmatory outcome

OTHER OUTCOMES:
Food cravings over the past week as measured by the COEQ (Three factors: craving control, craving for sweet foods, craving for savory foods) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Food cravings as measured by the General Food Cravings Questionnaire - Trait | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Explicit food liking measured during the Leeds Food Preference Task | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Eating behavior including cognitive restraint and dietary disinhibition (Eating Inventory) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Weight-related self-efficacy (WEL-short form) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Mood as assessed using the PHQ-9 | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Symptoms of disordered eating including clinician-rated binge eating frequency (sum of objective and subjective binge eating frequency) as assessed by the Eating Disorder Examination (EDE) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Self-reported loss-of-control eating (Loss of Control Eating Scale [LOCES]) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome
Drive for thinness (Eating Disorder Inventory [EDI]) | Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  S1: Supportive secondary outcome
Ratings of food palatability and of nausea, thirst, and wellbeing fasting and in the 4 hours after consuming the standard breakfast meal | S1: Change from baseline to weeks 20, 40, and 60, and measures at week 72; S2: Week 72 endpoint controlling for S1 baseline
  Exploratory outcome
Food addiction measured by Yale Food Addiction Scale | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Exploratory outcome
Body image satisfaction (Body Satisfaction Scale) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Exploratory outcome
Weight-related self stigmatization by the Weight Bias Internalization Scale | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Exploratory outcome
Body weight (kg) | S1: Change from baseline to weeks 20, 40, and 60; S2: Week 72 endpoint controlling for S1 baseline
  Supportive secondary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gordon K, Matthews A, Zeller MH, Lin J. Practical guidelines for eating disorder risk mitigation in patients undergoing obesity treatment for the pediatric provider. Curr Opin Pediatr. 2024 Aug 1;36(4):367-374. doi: 10.1097/MOP.0000000000001356. Epub 2024 Apr 5. PMID 38655793